CLINICAL TRIAL: NCT02199119
Title: Effect of Television Viewing During Exercise on Subjective Appetite, Satiation, and Food Intake in 9 to 14 Year Old Children
Brief Title: Effect of Television Viewing and Exercise on Appetite, Satiety, and Food Intake in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, Assistant Professor and Director, Food Intake Regulation & Satiety, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: REB 2013-120
Record Dates: First submitted 2014-07-20; First posted 2014-07-24 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Childhood Obesity
Keywords: children; television; exercise; food intake; appetite; satiation
MeSH Terms: conditions — Pediatric Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Experimental): Sitting quietly for 30 min No TV No exercise
  Interventions: Behavioral: Sitting quietly
- TV viewing only (Experimental): watching TV for 30 min
  Interventions: Behavioral: TV viewing
- Exercise only (Experimental): exercising for 30 min
  Interventions: Behavioral: Exercise
- TV viewing and Exercise (Experimental): 30 min of moderate exercise on a treadmill while watching TV
  Interventions: Behavioral: Exercise; Behavioral: TV viewing

INTERVENTIONS:
Behavioral: Exercise — 30 min of moderate exercise on a treadmill
  Arms: Exercise only; TV viewing and Exercise
Behavioral: TV viewing — watching TV (animated children's programming) for 30 min
  Arms: TV viewing and Exercise; TV viewing only
Behavioral: Sitting quietly — Sitting quietly for 30 min
  Arms: Control

SUMMARY:
The purpose of this study was to describe the effect of 30 min TV viewing with or without simultaneous moderate exercise using a treadmill on subsequent subjective appetite, satiation, and food intake in normal weight 9 to 14 year old children. It is hypothesized that TV viewing during exercise immediately before mealtime affects food intake regulation through its effect on the control of appetite and satiation.

ELIGIBILITY:
Inclusion Criteria:

* overall healthy, normal weight (between the 5th and 85th BMI percentile for age and gender) 9 to 14 year old boys and girls (peripubertal) born at term and at a normal birth weight, and does not receive any medications

Exclusion Criteria:

* significant learning, behavioral, or emotional difficulties, restricted diet, food allergies to test treatments

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Food Intake kcal | 30 min after end of treatment
  food is weighed pre and post consumption

SECONDARY OUTCOMES:
Subjective appetite and satiation in mm | measured at time 0, 15, 30, and 60 min
  Subjective appetite determined by visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Nick Bellissimo, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- FIRST Lab, Ryerson University, Toronto, Ontario, Canada